CLINICAL TRIAL: NCT01552382
Title: Vitamin D and Clinical Outcome in Cardiac Surgical Patients
Brief Title: Vitamin D, Cardiac Surgery and Outcome
Acronym: Vitop
Status: Completed | Type: Observational
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Sponsor
Other Study IDs: 006
Record Dates: First submitted 2012-02-07; First posted 2012-03-13 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2013-12

CONDITIONS: Cardiovascular Disease
Keywords: vitamin D; 25-hydroxyvitamin D; MACCE; mortality; cardiac; cerebrovascular
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cardiac surgical patients: patients undergoing a cardiac surgical procedure

SUMMARY:
We will use a retrospective data analysis to evaluate the association of vitamin D status with clinical outcome in cardiac surgical patients. The occurrence of several postoperative adverse events such as myocardial infarction, low cardiac output syndrome, stroke and in-hospital death will be assessed from cardiac surgery to discharge. In addition, we will assess the association of vitamin D status with the duration of mechanical ventilatory support and intensive care unit stay from cardiac surgery to discharge. Moreover, in-hospital stay will be assessed according to vitamin D status.

DETAILED DESCRIPTION:
In a retrospective data analysis, we will evaluate the association of vitamin D status (circulating 25-hydroxyvitamin D) with MACCE (major cardiac or cerebrovascular event) in cardiac surgical patients. The occurrence of several postoperative adverse events such as myocardial infarction, low cardiac output syndrome, stroke and in-hospital death will be assessed from cardiac surgery to discharge. Approximately 4,500 data sets from January 2010 until the end of 2011 will be analyzed.In all patients, we will also assess the association of vitamin D status with the duration of mechanical ventilatory support and intensive care unit stay from cardiac surgery to discharge. Moreover, in-hospital stay will be assessed according to vitamin D status.

ELIGIBILITY:
Inclusion Criteria:

* cardiac surgical patients aged 18 years and older

Exclusion Criteria:

* age < 18 years
* heart transplant recipients
* pacemaker or defibrillator implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cardiac surgical patients
Sampling Method: Probability Sample
Enrollment: 4418 (Actual)
Dates: Start 2012-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
major cardiac or cerebrovascular event (MACCE) | Patients will be followed for an average time of 14 days from cardiac surgery to discharge
  MACCE is defined as in-hospital death, myocardial infarction, low cardiac output syndrome or stroke.

SECONDARY OUTCOMES:
duration of ventilatory support | Patients will be followed for an average time of 14 days from cardiac surgery to discharge
intensive care unit stay | Patients will be followed for an average time of 14 days from cardiac surgery to discharge
in-hospital stay | Patients will be followed for an average time of 14 days from cardiac surgery to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Armin Zittermann, PhD, Principal Investigator — Georgstrasse 11, 32545 Bad Oenyhausen, Heart Center NRW, Ruhr University Bochum
Locations (2):
- Germany (2):
  - Heart and Diabetes Center NRW, Bad Oeynhausen, North Rhine-Westphalia
  - Heart Center North Rhine-Westphalia, Bad Oeynhausen, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zittermann A, Kuhn J, Dreier J, Knabbe C, Gummert JF, Borgermann J. Vitamin D status and the risk of major adverse cardiac and cerebrovascular events in cardiac surgery. Eur Heart J. 2013 May;34(18):1358-64. doi: 10.1093/eurheartj/ehs468. Epub 2013 Jan 12. PMID 23315905